CLINICAL TRIAL: NCT03830827
Title: Efficacy of Mindfulness-based Relapse Prevention With or Without Vortioxetine on the Prevention of Relapse in Chronic Methamphetamine Users
Brief Title: MBRP + Vortioxetine VS MBRP on Preventing Relapse in Chronic MA Users
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Shenzhen Mental Health Center (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Attending Psychiatrist, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2018008
Record Dates: First submitted 2019-01-14; First posted 2019-02-05 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Relapse; Cognitive Impairment; Depression
MeSH Terms: conditions — Recurrence; Cognitive Dysfunction; Depression | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRP+vortioxetine intervention (Experimental): Participants who allocate to the experimental group will receive 8-week 10-20mg/day vortioxetine combined with MBRP intervention.The MBRP intervention is composed of 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists to prevent MA relapse.
  10-20mg/day vortioxetine will sent every day and 2-hour MBRP intervention per week until the end of 8-week intervention . They will also receive 10 visits: visit 1 (week 0): medical and psychiatric screening; visit 2-9 (week 1, 2, 3, 4, 5, 6, 7 and 8): depressive symptoms and cognitive function, MA use, and MA craving; visit 10 (week 24): MA use (assessment of relapse rates), assessment of depressive symptoms, improvement in cognition and MA craving.
  Interventions: Drug: Vortioxetine
- MBRP intervention (Experimental): Participants who allocate to the control group will receive 8-week 1-2#/day placebo combined with MBRP intervention.The MBRP intervention is composed of 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists to prevent MA relapse.
  1-2#/day placebo will sent every day and 2-hour MBRP intervention per week until the end of 8-week intervention . They will also receive 10 visits: visit 1 (week 0): medical and psychiatric screening; visit 2-9 (week 1, 2, 3, 4, 5, 6, 7 and 8): depressive symptoms and cognitive function, MA use, and MA craving; visit 10 (week 24): MA use (assessment of relapse rates), assessment of depressive symptoms, improvement in cognition and MA craving.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — 8-week 10-20mg/day vortioxetine; 2-hour MBRP intervention per week in 8 weeks
  Other Names: Mindfulness-based relapse prevention

SUMMARY:
This multicenter, double-blind, Randomized, parallel-group study in subjects with methamphetamine dependence was to assess the efficacy of MBRP combined with vortioxetine and MBRP alone on 24-week abstinence rates, improvement of cognition and depressive symptoms.

DETAILED DESCRIPTION:
Participants who allocate to the experimental group will receive 8-week 10-20mg/day vortioxetine combined with MBRP intervention. Participants who allocate to the control group will receive 8-week 1-2#/day placebo combined with MBRP intervention.

Vortioxetine (Brintellix®), a novel antidepressant for the treatment of adult with major depressive disorder, has been approved by the Chinese Food and Drug Administration in the use of China in 2018.

The MBRP intervention is composed of 8 weekly, 2-hour sessions delivered in small group format (10-14 participants) by two therapists to prevent MA relapse. In MBRP, therapists facilitate discussions and exercises and introduce the meditation practice component. Group sessions include discussions of mindfulness as a means of coping with MA craving, negative affect and painful cognitions/sensations that precipitate relapse, role-playing exercises, meditation practice and implement practice into high-risk situations and in daily life, as well as homework assignments.

Participants from both groups will also receive 10 visits: visit 1 (week 0): medical and psychiatric screening; visit 2-9 (week 1, 2, 3, 4, 5, 6, 7 and 8): depressive symptoms and cognitive function, MA use, and MA craving; visit 10 (week 24): MA use (assessment of relapse rates), assessment of depressive symptoms, improvement in cognition and MA craving.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-V diagnosis of MA dependence within the last year
2. completion or scheduled completion (i.e., within 2 weeks) of inpatient or intensive outpatient treatment for MA dependence.
3. express a wish to remain abstinent from MA use
4. be age 18 to 65
5. be fluent in speaking Mandarin and literate in Chinese and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of mindfulness techniques
6. willingness to randomization and attendance at treatment and assessment sessions
7. be able to attend all clinic visits without interruption
8. score greater than 16 on the HAM D17 and MADRS >= 26, as well as currently not on any psychotropics for treatment of depression

Exclusion Criteria:

1. Any current Axis I DSM-V psychiatric disorder other than MA or nicotine dependence that, in the clinician's opinion, warrants treatment or would preclude safe participation in the protocol, including, but not limited to: psychosis, schizophrenia, dementia, schizotypal personality disorder, borderline personality disorder, bipolar disorder, primary diagnosis of eating disorder, or chronic suicidality or homicidality, mental retardation et al.
2. Serious medical comorbidity requiring medical intervention or close supervision, including pacemakers, heart transplant, severe arrhythmias, or active atrial fibrillation, gross neurological disease
3. Suicide attempt in the last 3 months
4. Pregnant or breastfeeding women
5. Prior treatment with vortioxetine or already participated in the MBRP program
6. Fail to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
The Timeline Followback (TLFB) for MA relapse rates | 24 weeks
  The primary objective is Methamphetamine (MA) relapse rates will be assessed by the Timeline Follow Back (TFB) at weeks 1, 2, 3, 4, 5, 6, 7, 8, and 24. TLFB is a technique for assessing self-reported alcohol or drug consumption that can be used as a clinical and research tool to obtain a variety of quantitative estimates of MA use. This outcome measure integrates data from self-reported supplied in the Time Line Follow Back (a self-reported summary of all substance use over the previous week) with biological verification.

SECONDARY OUTCOMES:
Depressive symptoms will be assessed by Montgomery and Asberg Depression Rating Scale (MADRS, Chinese version) | 24 weeks
  The efficacy of intervention for depressive symptoms was measured by mean change in Montgomery-Asberg Depression Rating Scale (MADRS) depression score from Baseline (Visit 2) to Week 24 (Visit 10). MADRS is a 10-item rating scale designed to measure overall severity of the symptoms in depressive and to be sensitive to treatment effects. Symptoms are rated on a 7-point Likert scale from 0 (no symptom) to 6 (severe symptom) with an overall score range from 0 to 60. Participants were considered responsive to vortioxetine if their MADRS score decreased by 50% or more from baseline to the end of treatment，and to be in remission if their final MADRS score is less than 10. A higher score indicates a more severe symptom, and a lower score from the baseline indicates an improvement in symptoms.
Cognition function will be assessed by THINC-it® cognition screening tool | 24 weeks
  THINC-it® is a sensitive cognitive screening tool for measuring the change of cognitive function and determining whether cognitive function is impaired. It required approximately 10 to 15 minutes for administration. It includes variants of the Choice Reaction Time Identification Task (IDN), One-Back Test, Digit Symbol Substitution Test, Trail Making Test-Part B, and the Perceived Deficits Questionnaire for Depression-5-item (PDQ-5-D).

CONTACTS AND LOCATIONS:
Overall Officials: Yanhui Liao, MD, Principal Investigator — Sir Run Run Shaw Hospital

IPD SHARING:
Plan to Share IPD: Undecided